CLINICAL TRIAL: NCT06176209
Title: Validating a Brief Screening Tool With Biomarkers for Prediction of Chronic Post Traumatic Neck Pain: A Prospective Cohort Study
Brief Title: Validating a Brief Screening Tool With Biomarkers for Prediction of Chronic Post Traumatic Neck Pain
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Specialized Hospital for Polio and Accident Victims, Rødovre, Denmark (Unknown); Næstved-Slagelse-Ringsted Hospital Research Fund (Unknown); The Danish Victims Fund (Other Government); The Research and Implementation Unit PROgrez, Region Zealand,Denmark (Unknown)
Responsible Party: Principal Investigator, Christian Lynæs, PT MSc, University of Southern Denmark
Other Study IDs: 106498
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain Following Traffic Accident
Keywords: Heart rate variability; Hyperarousal; Whiplash; Posttraumatic Stress Symptom; Neck Pain; Biomarkers; Hair cortisol
MeSH Terms: conditions — Whiplash Injuries; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair Samples for analysis of cortisol prior to accident (i.e three month)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post traumatic neck pain (i.e. whiplash): To be considered eligible for inclusion participants must meet the following criteria:
  Inclusion criteria: 18-60 years of age, post-traumatic neck pain of a musculoskeletal nature without fractures or slippage of vertebrae acquired within the last 72 hours in connection an accident. Participants must be able to read and speak Danish.
  Exclusion criteria: Previous pain discomfort after similar accidents, existing chronic back pain at the time of the accident, diagnosed with concussion after the accident, suspected or known spinal pathology, including confirmed fracture or slippage of vertebrae at the time of the accident, previous back or neck surgery, spinal cord injuries, severe psychiatric history (e.g., schizophrenia and depression), trauma patients or existing rheumatological or neurological disorders.
  Interventions: Diagnostic Test: screening tool with biomarkers for prediction of chronic post traumatic neck pain

INTERVENTIONS:
Diagnostic Test: screening tool with biomarkers for prediction of chronic post traumatic neck pain — Diagnostic screening with biomarkers for prediction of chronic post traumatic neck pain

SUMMARY:
Early screening of posttraumatic neck pain after accidents

- A clinical prediction tool with biomarkers predicting chronic posttraumatic neck pain.

The goal of this prospective cohort study is to develop a clinical prediction tool with biomarkers for early prediction of chronic posttraumatic neck pain.

Aims:

1. validate and further develop an existing prediction and screening tool for post traumatic neck pain using biomarkers for stress (i.e. HRV). The investigators hypothesize that the addition of a HRV to the existing screening and prediction tool in the acute phase (i.e. < 72 hours) post-accident can contribute to better and earlier identification of high-risk patients who continue to experience moderate to high degree of impairment after 12 months (i.e. NDI >32%).
2. examine whether the health economic costs for the group that does not improve are greater after 12 months. The investigators hypothesize that the health economic costs for the group that does not improve are greater after 12 months (labour market attachment and health services) compared to those who improve (NDI score < 10% vs. > 32%).
3. evaluate the role of low HRV on the development of PTSD 3 month after the accident. the hypothesis is that low HRV is a predictor of the development of PTSD.3 month after an accident.
4. Evaluate whether PTSD mediates the association between low HRV and pain sensitization 3 months after the accident. The investigators hypothesize that the development of pain sensitivity 3 month after an accident is associated with low HRV and PTSD.

Following inclusion participants will undergo evaluation of:

Hart rate variability using Fristbeat Bodyguard II, neurologic screening, Cervical range of motion screening.

At followup (1- and 3-months) participants will undergo evaluation of. Evaluation of cervical range of motion, Quantitative sensory testing (pressure pain threshold, cold pressor test followed by pressure pain threshold.

Questionnaires: Acute self-reported stress (NRS), Expected improvement (0-100%), Pain (Short Form -McGill pain questionnaire) Neck disability index, Stress, anxiety and depression, post-traumatic stress disorder, Pain catastrophizing, Quality of life, Global rating of change, Self-reported sleep, Comorbidity, Physical Activity.

At 6- and 12- month: Evaluation of heart rate variability and the questionnaires from 1- week and 3 months will be repeated.

DETAILED DESCRIPTION:
Background Post-traumatic neck pain sustained after accidents are frequent (1) and represents a huge human and societal burden that can cause significant long-term pain and disability (2-4). It has been estimated that there are 6,000 new annual cases of traffic accidents resulting in post-traumatic neck pain in Denmark (5). However, recent international research indicates that the figure may be more than double (6-8). While up to half of those injured continue to experience symptoms a year after the accident (1-3), 15-25% experience significantly more severe symptoms and functional impairment (9,10) and are at risk of leaving the labour market. The accumulated cost of post traumatic neck pain in Denmark has not been evaluated in a scientific study but it is estimated the direct and indirect economic costs of post traumatic neck pain are approximately DKK 14 billion annually (11).

Post-traumatic neck pain after accident is often accompanied by a myriad of symptoms such as headaches, fatigue, concentration problems, and sensitivity to light and sound (4,12-16). A number of studies also point to frequent psychological symptoms after injuries such as symptoms of stress, depression, and anxiety (15-17), and early post-traumatic stress has been reported to predict poorer recovery over time (18,19).

Previous studies have identified the same risk factors after whiplash injuries (20-26). Risk factors are age, high pain intensity, hypersensitivity to pain, and post-traumatic arousal symptoms (i.e. increased stress) immediately after the accident. The results suggest that the lack of efficacy of existing treatments (27-30) :is caused by not specifically targeting risk patients and the underlying related mechanisms.

Ritchie and colleagues have developed and validated a clinical prognostic screening tool to identify patients at risk of developing post traumatic neck pain (31,32). The optimal use of the screening tool is immediately after accidents. Based on simple screening questions that can be answered in less than 5 minutes regarding pain and related functional limitations, post-traumatic stress disorder (hyperarousal) and age, the screening tool can with 90% accuracy be used to identify those that do not improve after the accident and with 80% accuracy those who recovers completely. However, there is a need to test the screening tool in a Danish context in the emergency department and investigate whether biomarkers for stress can improve the predictive value of the tool.

In Denmark, the standard emergency department treatment after non traumatic accident is a thorough physical evaluation coupled with good advice, which is appropriate for a significant proportion of patients. Unfortunately, it is difficult to distinguish a normal reaction from a treatment-requiring reaction, which in turn can lead to a worsening of traumatic neck pain. In this instance the prognostic tool (31,32) will be simple and quick to use. Collection of objective biomarkers for early stress response immediately after the accident will probably strengthen the value of the tool and provide more insight into causal mechanisms in the development of chronic post-traumatic neck pain. Moreover, biomarkers such as heart rate variability (HRV) can be collected immediately after an accident and thereby predict the risk of developing PTSD. Using questionnaires this information would take weeks to collect risking delayed identification of risk patients.

A significant and recurring finding is that stress response immediately after an accident is a significant factor in the development of chronic post-traumatic neck pain. Post-traumatic arousal is associated with increased sensitivity to pain, catastrophic thinking, and misinterpretation of common bodily symptoms (33,34). An important biomarker for autonomic dysregulation (stress response) and development of post-traumatic stress symptoms is low HRV accompanied by high resting heart rate (35-41). Conversely, a high HRV is associated with cardiovascular recovery and improved self-regulation during stressful situations (42). To the best of our knowledge, only one study examined HRV as a predictor of PTSD after severe traffic trauma and found that HRV measured two days after an accident correctly identified 72% of those who developed PTSD after the accident (43).

Questionnaires Participants will be asked to answer questionnaires regarding quality of life, sleep, comorbidities, PTSD symptoms and physical activity. All questionnaires are validated in Danish. Questionnaires will be pilot tested at both sites before given to participants. Time consumption is estimated to 30 minutes and will be completed using a tablet when attending the emergency department and online during follow-up at 6 and 12 months respectively.

Clinical assessment The study uses a combination of different measurements such as self-reported variables, biomarkers (HRV), pain sensitivity tests (QST) and register data. Data will be collected at different time points.

During the initial visit in the emergency department a clinical assessment of the participants active range of motion of the cervical spine and upper and lower limbs will be conducted. Any pain, restriction in range of motion or discomfort will be noted. A complete neurological assessment of the upper and lower extremities will be performed. Isometric muscle strength and tendon reflexes will also be assessed. The clinical assessment including measurements of range of motion will be repeated during the follow up visit 1 week after the accident.

HRV HRV, resting heart rate, respiration frequency and sleep patterns form the study's biomarker for stress and are measured with the Firstbeat Bodyguard 2 tracker (Firstbeat Technologies Ltd., Finland) which records data continuously over four days. Measurements of HRV will be carried out at baseline, 3,6,12 month. HRV measurements can be used as a measurement of stress and recovery (45).

Quantitative sensory testing

The investigators l perform pressure pain thresholds and conditioned pain modulation at baseline and 3 month. Conditioned pain modulation will consist of pressure pain threshold followed by cold pressor test and pressure pain threshold. Pressure pain threshold will be performed in the lower limb (upper anterolateral aspect of the tibia). Immediately after the pressure pain threshold test participants will be asked to submerge their non-dominant hand in 0-2 degrees cold water for a maximum of 2 minutes or until pain is intolerable. Immediately here after the pressure pain threshold will be performed once again. Pressure pain threshold will be measured using an algometer (Somedic, Sweden). QST will be carried out on the non-dominant side. The protocol for QST will conform to the German Network for Neuropathic Pain protocol (46).

Follow up at 3, 6, and 12 months The participants will be contacted by phone at 3, 6 and 12 months. At 3 months another appointment for onsite testing will be arranged. At 6 and 12 months the FirstBeat device will be sent to participants by mail and participants will be asked to repeat the previous questionnaires online.

Sample size calculation and statistical analysis plan Based on previous cohort studies, it is expected that at least 25% of the participants will develop moderate to severe chronic symptoms (20,21,23,24,26). A more conservative estimate of 15% is used as the starting point for power calculation (easyROC web-tool v1.3.1). At an expected AUC of 0.80 and an allocation ratio of 7, a sample of 104 patients will be sufficient to give a statistical strength of 90% and yield a significant result (alpha 0.01). Drop-out rates and missing data are expected, hence an expected drop-out rate at 12-month follow-up of up to 25% is estimated. Thus, a total of 155 patients will be included. Distribution of normality will be examined using histogram and qq-plots. Parametric and non-parametric analysis will be applied as applicable. Participants' characteristics will be described at all time points.

The prediction tool will be validated by analysing its ability to predict those who recover from the traffic accident (NDI < 10%) and those who develop moderate to severe symptoms (NDI > 32%) at 12 months follow-up. The precision of the tool will be examined with receiver operator characteristics (ROC) analysis, and sensitivity and specificity are calculated by various cut-off criteria. In addition, logistic regressions will be performed as applicable with and without biomarkers in order to establish the best prediction model. Health economic costs are compared between groups. Labour market attachment, consumption of medicines and health services will serve as a proxy of recovery after 12 months for the groups identified by the prediction tool. All register data will be collected after 12-month follow-up has ended for all participants.

A multivariable regression analysis will be used to investigate the association between PTSD and HRV and participant data adjusted for relevant cofounders. Relevant confounders will be identified using directed acyclic graph (DAG)(47) specifically the dagitty tool for R package (48). Missing data will be managed by applying multiple imputation strategies. All data will be analysed using Stata (V.17, StataCorp, Texas, USA) and R (version 4.3.1 (Beagle Scouts)). The result of the analysis will be reported in accordance with STROBE statement (49) for cohort studies.

Ethics and dissemination The study is approved by the regional Ethics Committee (S-20230037) and the University of Southern Denmark, the study will also be registered at ClinicalTrials.gov. The study will conform with GDPR and the Data Protection Act as well as the declaration of Helsinki (50,51). Access to register data will be applied for via Statistics Denmark. Adverse events (AE) will be reported according to the regional Ethics Committee. Furthermore, AE will be recorded at all follow-up visits by asking participants about potential AEs using open questions to make sure all AEs are recorded. An AE is defined as any unwanted experience during follow-up leading to interaction with the healthcare system (General practitioner or hospital) due to symptom worsening.

Apart from possible short term pain flare up following the QST procedure there are no known significant long-term side effects of the data collection process. The design of this study does not allow for the minimum requirement of 24 hours of reflection time for participants. This procedure has been used before in the emergency department, and the procedure is approved by the regional Ethics Committee.

The results of the project will be published in peer-reviewed scientific journals as well as non-scientific dissemination in the form of articles in patient and professional journals and through press releases and social media. Practical workshops will be held to train interested professionals in the screening method - should this prove useful and effective. The result of this project will be published regardless of the magnitude or direction of the result. Co-authorships will be based on the ICMJE recommendations (52).

Perspectives and implications The results of this study should be of interest to clinicians, researchers, legal and insurance companies and policymakers and will strengthen both national and international knowledge about early identification of patients in high risk of developing chronic neck pain and the role of biomarkers. To our knowledge, this project is the first of its kind in a European context. If the findings of this study are positive, the investigators expect it will allow us to target resources more efficient and possibly cut the human cost of post traumatic neck pain.

Funding The project has received financial support from the University of Southern Denmark, and the Næstved-Slagelse-Ringsted Hospital Research Fund. None of the funders of this project will have influence on whether and how results are published, just as funders will have no influence on the choice of research design, content and the preparation of this protocol.

"These materials have received financial support from The Danish Victims Fund The execution, content, and results of the materials are the sole responsibility of the authors. The analysis and viewpoints that have been made evident form the materials belong to the authors and do not necessarily reflect the views of The Council of The Danish Victims Fund".

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* post-traumatic neck pain of a musculoskeletal nature without fractures or slippage of vertebrae acquired within the last 72 hours after accident.
* Participants must be able to read and speak Danish

Exclusion Criteria:

* Existing chronic pain at the time of the accident
* Suspected or known spinal pathology, including confirmed fracture or slippage of vertebrae at the time of the accident
* Previous back or neck surgery
* Spinal cord injuries
* Severe psychiatric history (e.g., schizophrenia and depression)
* Existing rheumatological or neurological disorders

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Participants presenting with neck pain after an accident
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | 72 hours after accident
  Neck pain and disability
Neck disability index | 1 week after accident
  Neck pain and disability
Neck disability index | 3 month after accident
  Neck pain and disability
Neck disability index | 6 month after accident
  Neck disability index
Neck disability index | 12 month after accident
  Neck disability index

SECONDARY OUTCOMES:
Heart Rrate Variability, respiration frequency, resting heart rate and sleep | <72 hours after accident
  Heart Rrate Variability, respiration frequency, resting heart rate and sleep measured with FirstBeat Bodyguard II
Heart Rrate Variability, respiration frequency, resting heart rate and sleep | 3 moths after accident
  Heart Rrate Variability, respiration frequency, resting heart rate and sleep measured with FirstBeat Bodyguard II
Heart Rrate Variability, respiration frequency, resting heart rate and sleep | 6 moths after accident
  Heart Rrate Variability, respiration frequency, resting heart rate and sleep measured with FirstBeat Bodyguard II
Heart Rrate Variability, respiration frequency, resting heart rate and sleep | 12 moths after accident
  Heart Rrate Variability, respiration frequency, resting heart rate and sleep measured with FirstBeat Bodyguard II
Neck mobility | < 72 hours after accident
  Neck mobility measured using a digital goniometer
Neck rotation | 1 week after accident
  Neck mobility measured using a digital goniometer
Neck rotation (CROM) | 3 month after accident
  Neck mobility measured using a digital goniometer
neurological evaluation | < 72 hours after accident
  neurological evaluation of force (grade 1-5) sensibility and reflexes in arms and legs
neurological evaluation | 1 week after accident
  neurological evaluation of force (grade 1-5) sensibility and reflexes in arms and legs
neurological evaluation | 3 month after accident
  neurological evaluation of force (grade 1-5) sensibility and reflexes in arms and legs
Pain sensitivity (QST) | 1 week after accident
  Pressure pain threshold followed by cold pressor test followed by pressure pain threshold
Pain sensitivity (QST) | 3 month after accident
  Pressure pain threshold followed by cold pressor test followed by pressure pain threshold
Acute self-reported stress (NRS) | < 72 hours after accident
  Acute self-reported stress (NRS)
Acute self-reported stress (NRS) | 1 week
  Acute self-reported stress (NRS)
Acute self-reported stress (NRS) | 3 month after accident
  Acute self-reported stress (NRS)
Acute self-reported stress (NRS) | 6 month after accident
  Acute self-reported stress (NRS)
Acute self-reported stress (NRS) | 12 month after accident
  Acute self-reported stress (NRS)
Patient Expected improvement (0-100%) | < 72 hours after accident
  Patient Expected improvement (0-100%)
Patient Expected improvement (0-100%) | 1 week after accident
  Patient Expected improvement (0-100%)
Patient Expected improvement (0-100%) | 3 month after accident
  Patient Expected improvement (0-100%)
Patient Expected improvement (0-100%) | 6 month after accident
  Patient Expected improvement (0-100%)
Patient Expected improvement (0-100%) | 12 month after accident
  Patient Expected improvement (0-100%)
Pain (SF-MPQ) | 1 week after accident
  Distribution of pain as evaluated by the SF (MPQ)
Pain (SF-MPQ) | 3 month after accident
  Distribution of pain as evaluated by the SF (MPQ)
Pain (SF-MPQ) | 6 month after accident
  Distribution of pain as evaluated by the SF (MPQ)
Pain (SF-MPQ) | 12 month after accident
  Distribution of pain as evaluated by the SF (MPQ)
Level of function (NDI) | 1 week after accident
  Level of function (NDI) instruments form the Neck disability index
Level of function (NDI) | 3 month after accident
  Level of function (NDI) instruments form the Neck disability index
Level of function (NDI) | 6 month after accident
  Level of function (NDI) instruments form the Neck disability index
Level of function (NDI) | 12 month after accident
  Level of function (NDI) instruments form the Neck disability index
Stress, anxiety and depression (DASS-21) | 1 week after accident
  Stress, anxiety and depression (DASS-21)
Stress, anxiety and depression (DASS-21) | 3 month after accident
  Stress, anxiety and depression (DASS-21)
Stress, anxiety and depression (DASS-21) | 6 month after accident
  Stress, anxiety and depression (DASS-21)
Stress, anxiety and depression (DASS-21) | 12 month after accident
  Stress, anxiety and depression (DASS-21)
PTSD (PDS, PCL-5) | 1 week after accident
  PTSD (PDS, PCL-5)
PTSD (PDS, PCL-5) | 3 month after accident
  PTSD (PDS, PCL-5)
PTSD (PDS, PCL-5) | 6 month after accident
  PTSD (PDS, PCL-5)
PTSD (PDS, PCL-5) | 12 month after accident
  PTSD (PDS, PCL-5)
Pain catastrophizing (PCS) | 1 week after accident
  Pain catastrophizing (PCS)
Pain catastrophizing (PCS) | 3 month after accident
  Pain catastrophizing (PCS)
Pain catastrophizing (PCS) | 6 month after accident
  Pain catastrophizing (PCS)
Pain catastrophizing (PCS) | 12 month after accident
  Pain catastrophizing (PCS)
Quality of life (EQ-5D-5L) | 1 week after accident
  Quality of life (EQ-5D-5L)
Quality of life (EQ-5D-5L) | 3 month after accident
  Quality of life (EQ-5D-5L)
Quality of life (EQ-5D-5L) | 6 month after accident
  Quality of life (EQ-5D-5L)
Quality of life (EQ-5D-5L) | 12 month after accident
  Quality of life (EQ-5D-5L)
Global rating of change (PGIC) | 1 week after accident
  Global rating of change (PGIC)
Global rating of change (PGIC) | 3 month accident
  Global rating of change (PGIC)
Global rating of change (PGIC) | 6 month accident
  Global rating of change (PGIC)
Global rating of change (PGIC) | 12 month accident
  Global rating of change (PGIC)
Self-reported sleep (KSS) | 1 week after accident
  Self-reported sleep (KSS)
Self-reported sleep (KSS) | 3 month after accident
  Self-reported sleep (KSS)
Self-reported sleep (KSS) | 6 month after accident
  Self-reported sleep (KSS)
Self-reported sleep (KSS) | 12 month after accident
  Self-reported sleep (KSS)
Comorbidity (GLA:D) | 1 week after accident
  Comorbidity (GLA:D)
Comorbidity (GLA:D) | 3 month after accident
  Comorbidity (GLA:D)
Comorbidity (GLA:D) | 6 month after accident
  Comorbidity (GLA:D)
Comorbidity (GLA:D) | 12 month after accident
  Comorbidity (GLA:D)
Physical Activity (GLA:D) | 1 week after accident
  Self reported Physical Activity (GLA:D)
Physical Activity (GLA:D) | 3 month after accident
  Self reported Physical Activity (GLA:D)
Physical Activity (GLA:D) | 6 month after accident
  Self reported Physical Activity (GLA:D)
Physical Activity (GLA:D) | 12 month after accident
  Self reported Physical Activity (GLA:D)

OTHER OUTCOMES:
DREAM | 24 month after accident
  registry data from The register-based evaluation of the extent of marginalization in Denmark
The National Patient Register | 24 month after accident
  Information about the use of health services for individual participants
The Register of Pharmaceutical Sales | 24 month after accident
  Information about the use of Pharmaceutical intervention for individual participants

IPD SHARING:
Plan to Share IPD: No
Not shared

REFERENCES:
- [Derived] Lynaes C, Ravn SL, Skou ST, Mogensen CB, Arvig MD, Christensen SWM, Sterling M, Andersen TE. Long-term recovery from post-traumatic neck pain: protocol for a prospective cohort study in the emergency department. BMJ Open. 2025 Nov 21;15(11):e099236. doi: 10.1136/bmjopen-2025-099236. PMID 41271421